CLINICAL TRIAL: NCT00437281
Title: A Placebo-Controlled, Escalating Dose, Multiple Dose Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Pregabalin In Pediatric Patients With Partial Onset Seizures
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of Pregabalin in Pediatric Patients With Partial Onset Seizures
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081074
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2014-01

CONDITIONS: Epilepsies, Partial
Keywords: Partial-onset seizures; epilepsy; pediatric; pregabalin; safety; tolerability; pharmacokinetics
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Pregabalin — Orally-administered pregabalin
  Arms: Pregabalin

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of multiple doses of pregabalin in pediatric patients with partial onset seizures that are incompletely controlled on their current medications.

ELIGIBILITY:
Inclusion Criteria:

* Partial onset seizures, incompletely controlled on 1-3 medications
* At least 1 seizure per 28 days, on average

Exclusion Criteria:

* Primary generalized seizures
* Progressive CNS pathology

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2007-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (13):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Gulf Breeze, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
- Mexico (2):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- [Derived] Mann D, Liu J, Chew ML, Bockbrader H, Alvey CW, Zegarac E, Pellock J, Pitman VW. Safety, tolerability, and pharmacokinetics of pregabalin in children with refractory partial seizures: a phase 1, randomized controlled study. Epilepsia. 2014 Dec;55(12):1934-43. doi: 10.1111/epi.12830. Epub 2014 Nov 6. PMID 25377429
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081074&StudyName=Safety%2C%20Tolerability%2C%20and%20Pharmacokinetic%20Study%20of%20Pregabalin%20in%20Pediatric%20Patients%20with%20Partial%20Onset%20Seizures

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed this study and who tolerated study medication were eligible to enroll in study A0081075 (NCT00448916), a 12-month open-label extension study of pregabalin.
Groups:
- Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received pregabalin oral liquid formulation 2.5 milligram per kilogram per day (mg/kg/day) in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received pregabalin oral liquid formulation 5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received pregabalin oral liquid formulation 10 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received pregabalin oral liquid formulation 15 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg, 2.5 mg/kg, 5 mg/kg or 7.5mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received pregabalin oral liquid formulation 2.5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received pregabalin oral liquid formulation 5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received pregabalin oral liquid formulation 10 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received pregabalin oral liquid formulation 15 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg, 2.5 mg/kg, 5 mg/kg or 7.5mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received pregabalin oral liquid formulation 2.5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received pregabalin oral liquid formulation 5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received pregabalin oral capsule 10 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received pregabalin oral capsule 15 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received placebo matched to pregabalin oral liquid formulation or capsule 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg or 2.5 mg/kg, or pregabalin oral capsule 5 mg/kg or 7.5mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received pregabalin oral liquid formulation 2.5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received pregabalin oral liquid formulation 5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received pregabalin oral capsule 10 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received pregabalin oral capsule 15 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received placebo matched to pregabalin oral liquid formulation or capsule 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg or 2.5 mg/kg, or pregabalin oral capsule 5 mg/kg or 7.5mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
Period: Overall Study
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Placebo (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Placebo (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Placebo (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) | Placebo (Age Cohort: 12 to 16 Years)
Started | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 3 | 5 | 3 | 3 | 4 | 2 | 3
Completed | 3 | 3 | 3 | 2 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 2 | 4 | 3 | 3 | 4 | 1 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Placebo (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Placebo (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Placebo (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) | Placebo (Age Cohort: 12 to 16 Years) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 3 | 5 | 3 | 3 | 4 | 2 | 3 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.2 (0.7) | 1.4 (0.5) | 0.7 (0.5) | 0.6 (0.1) | 1.6 (0.3) | 4.0 (0.8) | 2.9 (0.1) | 4.0 (1.7) | 3.9 (1.8) | 3.7 (1.0) | 9.3 (1.2) | 9.7 (2.3) | 10.0 (0.0) | 9.0 (1.0) | 9.2 (1.5) | 15.7 (0.6) | 13.7 (2.1) | 14.0 (1.8) | 15.5 (0.7) | 13.0 (1.7) | 6.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 2 | 4 | 2 | 1 | 1 | 3 | 2 | 1 | 0 | 0 | 4 | 2 | 1 | 0 | 0 | 3 | 32
  Male | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 3 | 1 | 1 | 2 | 4 | 2 | 0 | 33

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Clinically Significant Change in Physical and Neurological Findings
Description: Full physical examination included examination of the abdomen, breasts, lungs, lymph nodes, mouth, genitourinary, musculoskeletal and neurological systems, skin, extremities, head, heart, ears, eyes, neck, nose, ocular fundi, throat and thyroid gland. The neurological exam was performed by a pediatric neurologist or qualified investigator.
Time Frame: Baseline up to 7 days post-last dose of study medication
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Placebo (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Placebo (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Placebo (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) | Placebo (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 3 | 5 | 3 | 3 | 4 | 2 | 3
participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Treatment-Emergent Adverse Events (AEs) by Severity: Double-blind Treatment
Description: Analysis for severity of AEs was performed separately for double-blind and open-label treatment. AE = any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. AEs were classified as mild, moderate and severe based on severity assessment: Mild = no interference with participant's usual function; Moderate = some interference with participant's usual function; Severe = significant interference with participant's usual function. Treatment-emergent events for double-blind treatment included events between baseline and Day 7 that were absent before treatment or that worsened relative to pretreatment state. Participants may experience more than 1 AE.
Time Frame: Baseline to Day 7
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: adverse events
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Placebo (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Placebo (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Placebo (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) | Placebo (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 3 | 5 | 3 | 3 | 4 | 2 | 3
adverse events
  Mild | 0 | 2 | 2 | 4 | 1 | 1 | 4 | 5 | 5 | 13 | 0 | 3 | 3 | 5 | 2 | 0 | 2 | 11 | 2 | 0
  Moderate | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 4 | 3 | 0
  Severe | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0

3. Secondary Outcome: 28-Day Seizure Frequency Rate
Description: Seizure frequency was reported by participant's parent or guardian from randomization to 7 days post-last dose of study medication. 28-day seizure frequency rate = (number of seizures in observation period/number of days in observation period)*28.
Time Frame: Baseline up to 7 days post-last dose of study medication
Population: Results are not reported since the data was reported in individual participant listings but not summarized for analysis.
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Placebo (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Placebo (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Placebo (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) | Placebo (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau): Multiple-Dose Analysis
Description: Area under the curve from time zero to the end of dosing interval (AUCtau), where dosing interval was 12 hours, for participants who received pregabalin from Day 1 to Day 8 morning is reported (multiple-dose participants). Results are normalized to individual participant's Day 8 dose.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose on Day 8
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period (double-blind or open label treatment). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (microgram*hour/milliliter)/(mg/kg)
Groups:
- Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received pregabalin oral liquid formulation 2.5 mg/kg/day) in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 1 | 2 | 3 | 3 | 4 | 1
(microgram*hour/milliliter)/(mg/kg) | 7.614 (19) | 7.563 (26) | 7.595 (6) | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 7.962 (29) | NA (NA) — Geometric mean and coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | NA (NA) — Geometric mean and coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 8.203 (31) | 11.64 (29) | 9.571 (9) | 7.59 | NA (NA) — Geometric mean and coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 10.20 (13) | 13.07 (34) | 9.642 (44) | 14.4

5. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]: Single-Dose Analysis
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). AUC (0 - ∞) for participants who received matching placebo from Day 1 to Day 7 and pregabalin on Day 8 morning is reported (single-dose participants). Results are normalized to individual participant's Day 8 dose.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: PK parameter analysis population. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Results are not reported for pregabalin 10 and 15 mg/kg/day for 12 to 16 age cohort since none of the participant had PK parameter available in these groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (microgram*hour/milliliter)/(mg/kg)
Groups:
- Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 5 mg/kg (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 5 mg/kg (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 2 to 6 Years): Participants of 2 to 6 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 5 mg/kg (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received placebo matched to pregabalin oral capsule 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 7 to 11 Years): Participants of 7 to 11 years of age received placebo matched to pregabalin oral capsule 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received placebo matched to pregabalin oral liquid formulation 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 2.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 5 mg/kg (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received placebo matched to pregabalin oral capsule 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
- Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 12 to 16 Years): Participants of 12 to 16 years of age received placebo matched to pregabalin oral capsule 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral capsule 7.5 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
Arm/Group | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
(microgram*hour/milliliter)/(mg/kg) | 6.70 | 8.10 | 7.05 | 7.02 | 8.30 | 6.38 | 8.76 | 9.16 | 10.0 | 10.1 | 8.00 | 15.9 | 13.8 | 10.6 |  |

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): Multiple-Dose Analysis
Description: Cmax for participants who received pregabalin from Day 1 to Day 8 morning is reported (multiple-dose participants). Results are normalized to individual participant's Day 8 dose.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period (double-blind or open label treatment). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (microgram/milliliter)/(mg/kg)
Groups:
- Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months): Participants of 1 to 23 months of age received pregabalin oral liquid formulation 2.5 mg/kg/day in 2 equally divided doses 12 hours apart for 7 days as double-blind treatment. Single open-label morning dose of pregabalin oral liquid formulation 1.25 mg/kg on Day 8. Participants who discontinued or did not enter open-label extension study were tapered off medication over 1 week.
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 1 | 2 | 3 | 3 | 4 | 1
(microgram/milliliter)/(mg/kg) | 1.468 (23) | 1.577 (11) | 1.496 (14) | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 1.601 (13) | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 1.856 (15) | 2.350 (29) | 1.660 (13) | 0.945 | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 1.762 (22) | 2.538 (44) | 1.355 (59) | 1.94

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): Single-Dose Analysis
Description: Cmax for participants who received matching placebo from Day 1 to Day 7 and pregabalin on Day 8 morning is reported (single-dose participants). Results are normalized to individual participant's Day 8 dose.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (microgram/milliliter)/(mg/kg)
Arm/Group | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
(microgram/milliliter)/(mg/kg) | 1.51 | 1.81 | 1.18 | 1.52 | 1.93 | 1.50 | 1.70 | 1.54 | 1.31 | 2.29 | 1.24 | 1.28 | 1.81 | 1.79 |  |

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Multiple-Dose Analysis
Description: Tmax for participants who received pregabalin from Day 1 to Day 8 morning is reported (multiple-dose participants).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 1 | 2 | 3 | 3 | 4 | 1
hours | 0.617 [0.500 to 1.00] | 1.05 [1.00 to 2.08] | 1.12 [1.02 to 2.00] | 2.49 [0.967 to 4.02] | 0.500 [0.500 to 2.00] | 1.67 [1.17 to 2.17] | 2.62 [1.17 to 4.07] | 1.00 [0.967 to 1.17] | 0.583 [0.583 to 1.00] | 1.00 [1.00 to 1.00] | 4.00 | 0.790 [0.500 to 1.08] | 0.500 [0.500 to 4.00] | 0.583 [0.483 to 1.00] | 2.09 [1.50 to 8.08] | 2.15

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Single-Dose Analysis
Description: Tmax for participants who received matching placebo from Day 1 to Day 7 and pregabalin on Day 8 morning is reported (single-dose participants).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
hours | 1.00 | 0.967 | 1.13 | 1.00 | 0.450 | 1.00 | 1.00 | 1.98 | 1.00 | 0.583 | 2.00 | 4.00 | 4.05 | 1.00 |  |

10. Secondary Outcome: Plasma Decay Half-Life (t1/2): Multiple-Dose Analysis
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. t1/2 for participants who received pregabalin from Day 1 to Day 8 morning is reported (multiple-dose participants).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 1 | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 4 | 1
hours | 4.433 (0.17559) | 3.397 (0.58603) | 3.263 (0.49903) | NA (NA) — Arithmetic mean and standard deviation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 3.90 | NA (NA) — Arithmetic mean and standard deviation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 3.523 (0.25146) | 3.520 (0.91804) | 4.287 (0.27737) | 4.113 (0.25891) | NA (NA) — Arithmetic mean and standard deviation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | NA (NA) — Arithmetic mean and standard deviation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 4.960 (1.3857) | 3.953 (0.80532) | 5.643 (0.88921) | 6.61

11. Secondary Outcome: Plasma Decay Half-Life (t1/2): Single-Dose Analysis
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. t1/2 for participants who received matching placebo from Day 1 to Day 7 and pregabalin on Day 8 morning is reported (single-dose participants).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
hours | 2.64 | 3.78 | 3.76 | 3.22 | 3.88 | 2.70 | 3.83 | 3.08 | 4.77 | 4.02 | 3.13 | 6.54 | 5.80 | 3.85 |  |

12. Secondary Outcome: Apparent Oral Clearance (CL/F): Multiple-Dose Analysis
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed (F). Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F for participants who received pregabalin from Day 1 to Day 8 morning is reported (multiple-dose participants).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/minute (mL/min)
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 1 | 2 | 3 | 3 | 4 | 1
milliliter/minute (mL/min) | 19.00 (10) | 17.70 (47) | 18.54 (49) | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 34.18 (61) | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 30.49 (9) | 58.23 (42) | 49.49 (19) | 63.7 | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 90.56 (26) | 78.38 (12) | 85.87 (17) | 73.1

13. Secondary Outcome: Apparent Oral Clearance (CL/F): Single-Dose Analysis
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed (F). Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F for participants who received matching placebo from Day 1 to Day 7 and pregabalin on Day 8 morning is reported (single-dose participants).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
mL/min | 31.5 | 24.7 | 20.1 | 28.0 | 32.3 | 60.1 | 38.8 | 45.5 | 58.2 | 45.8 | 64.8 | 54.3 | 99.6 | 90.0 |  |

14. Secondary Outcome: Renal Clearance (CLr): Multiple-Dose Analysis
Description: Renal clearance is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time. CLr for participants who received pregabalin from Day 1 to Day 8 morning is reported (multiple-dose participants).
Time Frame: 0 to 12 hours post-dose, 12 to 24 hours post-dose on Day 8
Population: PK parameter analysis population. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Results are not reported for some of the groups since none of the participant had PK parameter available in these groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 2 | 3 | 0
mL/min |  | 21.0 |  |  | 8.77 |  | 48.4 | 11.5 |  | 24.75 (88) | 55.9 | 36.9 |  | NA (NA) — Geometric mean and geometric coefficient of variation obtained by sampling distribution of 2 participants were not considered meaningful, hence not analyzed. | 69.16 (39) |

15. Secondary Outcome: Renal Clearance (CLr): Single-Dose Analysis
Description: Renal clearance is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time. CLr for participants who received matching placebo from Day 1 to Day 7 and pregabalin on Day 8 morning was to be reported (single-dose participants).
Time Frame: 0 to 12 hours post-dose, 12 to 24 hours post-dose on Day 8
Population: PK parameter analysis population. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Results are only reported for pregabalin 15 mg/kg/day, 7 to 11 years and pregabalin 5 mg/kg/day, 12 to 16 years because none of the participant had PK parameter available in rest of the groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 1 to 23 Months) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 2 to 6 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 7 to 11 Years) | Placebo, Pregabalin 1.25 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 2.5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 5 mg/kg (Age Cohort: 12 to 16 Years) | Placebo, Pregabalin 7.5 mg/kg (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
mL/min |  |  |  |  |  |  |  |  |  |  |  | 42.6 |  | 73.8 |  |

16. Primary Outcome: Number of Treatment-Emergent Adverse Events (AEs) by Severity: Open-label Treatment
Description: Analysis for severity of AEs was performed separately for double-blind and open-label treatment. AE = any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. AEs were classified as mild, moderate and severe based on severity assessment: Mild = no interference with participant's usual function; Moderate = some interference with participant's usual function; Severe = significant interference with participant's usual function. Treatment-emergent events for open-label treatment included events between Day 8 and 28 days after the open-label dose that were absent before treatment or that worsened relative to pretreatment state. Participants may experience more than 1 AE.
Time Frame: Day 8 up to 28 days after open-label dose of study medication
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: adverse events
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Placebo (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Placebo (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Placebo (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) | Placebo (Age Cohort: 12 to 16 Years)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 3 | 5 | 3 | 3 | 4 | 2 | 3
adverse events
  Mild | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) | Placebo (Age Cohort: 1 to 23 Months) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) | Placebo (Age Cohort: 2 to 6 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) | Placebo (Age Cohort: 7 to 11 Years) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) | Placebo (Age Cohort: 12 to 16 Years)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/4 | 0/4 | 0/3 | 0/3 | 0/3 | 0/5 | 0/3 | 0/3 | 0/2 | 1/3 | 1/5 | 0/3 | 0/3 | 0/4 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/3 | 3/3 | 2/4 | 2/4 | 1/3 | 2/3 | 2/3 | 4/5 | 2/3 | 3/3 | 2/2 | 2/3 | 2/5 | 1/3 | 1/3 | 4/4 | 2/2 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Placebo (Age Cohort: 1 to 23 Months) (N=4) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=4) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=3) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=3) | Placebo (Age Cohort: 2 to 6 Years) (N=5) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=3) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=2) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=3) | Placebo (Age Cohort: 7 to 11 Years) (N=5) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=3) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=4) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=2) | Placebo (Age Cohort: 12 to 16 Years) (N=3)
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Pregabalin 5 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Pregabalin 15 mg/kg/Day (Age Cohort: 1 to 23 Months) (N=3) | Placebo (Age Cohort: 1 to 23 Months) (N=4) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=4) | Pregabalin 5 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=3) | Pregabalin 15 mg/kg/Day (Age Cohort: 2 to 6 Years) (N=3) | Placebo (Age Cohort: 2 to 6 Years) (N=5) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=3) | Pregabalin 5 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=2) | Pregabalin 15 mg/kg/Day (Age Cohort: 7 to 11 Years) (N=3) | Placebo (Age Cohort: 7 to 11 Years) (N=5) | Pregabalin 2.5 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=3) | Pregabalin 5 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=3) | Pregabalin 10 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=4) | Pregabalin 15 mg/kg/Day (Age Cohort: 12 to 16 Years) (N=2) | Placebo (Age Cohort: 12 to 16 Years) (N=3)
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tandem gait test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Learning disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Results are reported for AUCtau for multiple-dose PK analysis and AUC (0-∞) for single-dose PK analysis, instead of AUC (0-24), as per change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.